CLINICAL TRIAL: NCT07131852
Title: Structural Brain Volumetry Changes in Eating Disorders.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alya Mohamed, Assistant Lecturer, Assiut University
Other Study IDs: 645210
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Eating Disorders; Psychiatric Comorbidities
Keywords: Eating Disorders; Anorexia Nervosa; Binge eating disorders; bulimia disorders
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Binge-Eating Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Anorexia Nervosa Patients
- Bulimia Nervosa Patients
- Binge-Eating Disorder
- control group

SUMMARY:
The goal of this observational study is to investigate the relationship between structural brain changes and psychiatric comorbidities in individuals diagnosed with eating disorders (EDs). The main question it aims to answer is:

How are structural brain volumetric changes associated with psychiatric comorbidities in patients with eating disorders?

Participants with a clinical diagnosis of an eating disorder will undergo brain MRI scans for volumetric analysis and structured psychiatric assessments to identify comorbid conditions. Data will be collected cross-sectionally from patients receiving routine clinical care, with the aim of identifying neurobiological and psychiatric patterns that could inform targeted treatment and prevention strategies.

DETAILED DESCRIPTION:
Eating disorders (EDs) are complex psychiatric conditions characterized by persistent disturbances in eating behaviors, body weight regulation, and self-perception, often accompanied by severe physical health consequences and high mortality rates (1). They typically emerge during adolescence or early adulthood but may develop at any age, with a multifactorial etiology involving genetic, neurobiological, psychological, and sociocultural influences (2).

The main diagnostic categories include anorexia nervosa (AN)-marked by significantly low body weight, intense fear of weight gain, and body image distortion; bulimia nervosa (BN)-characterized by recurrent binge eating followed by compensatory behaviors such as vomiting, fasting, or excessive exercise; and binge-eating disorder (BED)-involving recurrent episodes of excessive food intake without compensatory behaviors (3). Other specified feeding or eating disorders (OSFED) encompass clinically significant presentations not meeting full criteria for the above disorders.

In Egypt, eating disorders represent an under-recognized public health concern. Recent epidemiological studies have found that approximately 13.3% of Egyptian youth meet criteria for an ED, with BN being the most prevalent (8.4%) and BED affecting 1.4% (4). The apparent absence of AN cases in some surveys may reflect cultural perceptions of thinness, under-diagnosis, and stigma rather than true absence (5). Risk factors identified in Egyptian samples include high body mass index (BMI), exposure to Westernized beauty ideals, depression, and a history of psychological trauma (6).

Structural neuroimaging, particularly MRI, has revealed consistent alterations in ED patients. AN is often associated with global and regional gray matter reductions-particularly in the parietal, frontal, and temporal cortices-along with decreased subcortical and cerebellar volumes (7). BN has been linked to structural changes in frontal and striatal regions, potentially reflecting alterations in impulse control and reward processing (8). Some volumetric changes may partially reverse with nutritional rehabilitation, suggesting neuroplasticity (9).

Psychiatric comorbidities are highly prevalent in EDs, affecting more than 70% of patients (10). Anxiety disorders, mood disorders, obsessive-compulsive disorder (OCD), post-traumatic stress disorder (PTSD), and substance use disorders are common, often worsening symptom severity and complicating treatment (10, 11). OCD traits are especially frequent in AN, while BN shows strong associations with depression and anxiety.

This study aims to use structural MRI to investigate brain volumetric changes in individuals with eating disorders and to explore the relationship between these changes and psychiatric comorbidities, thereby contributing to a more comprehensive understanding of the neuropsychiatric profile of EDs.

ELIGIBILITY:
Inclusion Criteria:

* Age above 13 years.
* DSM-5 diagnosis of an eating disorder (AN, BN, BED) confirmed by structured interview.

Exclusion Criteria:

* Neurological or any previous psychiatric diagnosis.
* IQ less than 70.
* MRI contraindication (metal implants, pacemaker, severe claustrophobia).

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study Setting: in Assuit university hospitals, Neuropsychiatry hospital Outpatient Clinic Study subjects: will include three groups of patients with eating disorders: Anorexia nervosa patients, Bulimia Nervosa patients, Binge-eating patients, and healthy control group they will be age and sex matched.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-02-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
To assess structural changes of brain volumetry in patients with eating disorders and compare with healthy controls. | from enrollment till 18 months

SECONDARY OUTCOMES:
Highlight the extent of psychological disorders in such patients. | From enrollment till 18 months

IPD SHARING:
Plan to Share IPD: Undecided